CLINICAL TRIAL: NCT03856177
Title: A Novel Bench-to-Bedside Translational Model of Anhedonia
Brief Title: Translational Model of Anhedonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Cavanagh, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R01MH119382-01 (NIH); 1R01MH119382-01 (NIH)
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into neutral or emotionally evocative conditions prior to assessing EEG brain signals of reward.
Who Masked: Investigator
Masking Description: Randomization will be based on the last digit (odd vs. even) of the participant's research identifier.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutral (Experimental): A neutral mood induction will include reading a dull text while listening to non-evocative music for 5-15 minutes.
  Interventions: Behavioral: Emotion Induction
- Evocative (Experimental): A mood induction procedure will be utilized. The procedure consists of a combination of re-experiencing an autobiographical sad personal event while listening to their choice of one of four sad music selections commonly used in mood induction. Visual analogue scale ratings will assess momentary sadness prior to, following, and at subsequent time points around the mood induction procedure.
  Interventions: Behavioral: Emotion Induction

INTERVENTIONS:
Behavioral: Emotion Induction — Described in arm

SUMMARY:
The proposed research addresses a major mental health issue (anhedonia) with a novel computationally-inspired translational technique in both humans and mice. This approach greatly increases the likelihood that a positive animal model result will be successfully translated to humans. This research plan thus offers a novel way to address the NIMH's mission of defining mechanisms of complex behaviors.

DETAILED DESCRIPTION:
Although considered a trans-diagnostic phenotype, anhedonia can emerge from deficits in motivation, valuation, or hedonic appreciation, each of which reflect different neural processes and are differently expressed across individuals. There is a critical need to refine the construct of anhedonia in order to improve treatment. The long-term goal of this project is to combine computational, imaging, and causal manipulations to define a translational biomarker of diminished valuation in anhedonia. This proposal aims to identify how the EEG response known as the Reward Positivity (RewP) is a candidate biomarker specific to value-based deficiencies in anhedonia. The RewP is only elicited by the presentation of a rewarding outcome, it is decreased in depression, and it scales with the central feature of reinforcement learning models, the positive reward prediction error (+RPE). Importantly, this same neural response can be elicited in rodents using the same learning task as in humans. The objective of this proposal is to test whether induced emotion, depressed mood, and learned helplessness (in mice) directly diminish +RPE coding in the RewP. The rationale for this approach is that electrophysiology is a highly promising tool for identifying mechanisms of complex behaviors and translating these mechanisms between species. Aim 1 will determine if induced emotion and +RPE have independent or interactive effects on the RewP. Aim 2 will recruit depressed participants and determine if anhedonia and +RPE have independent or interactive influences on the source-level generators underlying the RewP (using MEG). Aim 3 will use the same task in a mouse model with infralimbic recordings; this will then test the causal diminishment (learned helplessness) and recovery (fluoxetine) of this mechanism. This proposed research is innovative because it identifies a computational function tightly tied to a neural response that directly addresses the disease-specific phenotype in human patients and is capable of being assessed, manipulated, and recovered within a rodent model. This contribution is expected to be significant because it will advance a translational mechanism for deficient valuation in anhedonia. Upon completion of these aims, the expected outcome will validate the RewP as a sensitive and specific mechanism of aberrant valuation in anhedonia. In line with the Research Domain Criteria framework, the use of computational modeling will facilitate algorithmic contrasts between multiple sub-constructs of approach motivation in the positive valence systems domain. The translational computational psychiatry approach advanced here links circuit-level dysfunction, aberrant computations, and trans-diagnostic behavioral phenotype. The successful completion of the aims advanced here will create a highly promising path for combining these strengths into a computationally-inspired, mechanistically tested, translatable model of aberrant valuation in anhedonia. This novel candidate biomarker will be translatable between species and testable in an outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-55
* Free from psychoactive medication for at least 2 weeks

Exclusion Criteria:

* Participants unwilling or unable to give informed consent
* Presence of other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study
* History of psychosis
* Not fluent in English

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico - Logan hall, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were run in the Cognitive Rhythms and Computation Lab at UNM from 6/13/19 - 5/7/21
Pre-assignment Details: There are no significant events to describe between enrollment and assignment.
Period: Overall Study
Arm/Group | Neutral | Evocative
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy non-depressed individuals 18-55 years old.
Groups:
- Total: Total of all reporting groups
Arm/Group | Neutral | Evocative | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 8 | 11
  White | 36 | 30 | 66
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Reward Positivity Component of the Event-Related Electroencephalogram
Description: The Reward Positivity is a fronto-centrally located positive voltage burst recorded in the EEG from about 200-500 ms following the receipt of a reinforcing outcome (e.g. money, points). Higher voltages (more positive numbers) indicate a larger reward response.
Time Frame: There will only be one day session (on the date of the randomization) where the Reward Positivity amplitude is assessed
Measure: Mean (Standard Deviation); unit: Microvolts
Arm/Group | Neutral | Evocative
Number analyzed (Participants) | 50 | 50
Microvolts | 7.29 (3.78) | 9.23 (3.64)
Statistical Analysis 1: Comparison: Neutral vs Evocative; Test type: Other; p = .071, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on the single day of the study. (1 day period of time).
Arm/Group | Neutral | Evocative
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03856177/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03856177/SAP_001.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03856177/ICF_002.pdf